CLINICAL TRIAL: NCT02789943
Title: The National Heart Centre Singapore Prospective CABG Cohort: Multi- Level and Integrated Analysis of Mechanisms Underlying Atrial Dysfunction
Brief Title: Multi- Level and Integrated Analysis of Mechanisms Underlying Atrial Dysfunction
Acronym: STaR-CABG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Heart Centre Singapore (Other)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/103/C
Record Dates: First submitted 2016-05-30; First posted 2016-06-03 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2016-05

CONDITIONS: Ischemic Heart Disease
Keywords: IHD Normal EF
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Tissue samples ( Atrial Appendage Tissue/ Aortic Button ) Blood Serum
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Cardiac Bypass Surgery — elective cardiac bypass surgery during which a sample of right atrial appendage and/ or aortic button can be removed

SUMMARY:
Integrated and cross-disciplinary analysis of human physiology and disease provides unbiased and deeply informative insights into human health and disease. In this study the investigators will recruit patients undergoing coronary artery bypass surgery to study the atrium of the heart or the aortic wall that when diseased can cause strokes.

Hypothesis: Systems-level analysis of the left atrium and aorta cells that integrates imaging, histological, cellular and molecular data will identify new mechanism for cardiovascular form and function.

DETAILED DESCRIPTION:
While there are many sub-aims to this study, the overarching goal is to define molecular mechanisms underlying atrial dysfunction. Here the investigator provide a power calculation based on detecting the genetic control points of gene expression (eQTLs) in the human atrial fibroblast. The investigator and many others have shown that tissue-specific eQTLs can be robustly identified at genome-wide significance in segregating populations of ~200. In this study the investigator propose eQTL association analysis in humans, which have previously been successfully performed in cohorts of less than 1000 subjects. The general applicability of this approach has been validated in multiple studies across multiple tissues in cohorts of between 200-1000 subjects.Based on published imaging genetic studies that have been successfully applied in small cohorts (<500) and the success of echo-based, semi-quantitative studies of ventricular dimensions, the investigator are confident that our quantitative studies of 750 individuals are powered to detect genome wide significant loci for the traits under study.

Despite intensive research there is a critical gap in our knowledge in the mechanisms underlying atrial fibrillation, which is a major cause of stroke and heart failure and increasingly common as it is a disease of the elderly. This project will address this important gap in our knowledge and provide new insights into disease pathogenesis with the goal of stratifying participants to prevent strokes and for treating the underlying substrate.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective cardiac bypass surgery during which a sample of right atrial appendage and/or aortic button can be removed.

Exclusion Criteria:

* Infection within 2 weeks preceding the operation or immunosuppressive therapy.
* Patients not able or willing to consent for study.
* Previous atrial intervention.
* Patients who cannot be followed up.
* Exclude patients with significant valvular disease (any planned valvular surgery, MR > severe, AS > severe, TR > severe).

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from wards or referral from clinics at the National Heart Centre Singapore if criteria is fulfil
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2013-05; Primary Completion 2017-07 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
First occurrence of cardiovascular event | One year

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Alexander Cook, Principal Investigator — National Heart Centre Singapore / Duke NUS Graduate Medical School
Locations (1):
- National Heart Centre, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hogue CW Jr, Creswell LL, Gutterman DD, Fleisher LA; American College of Chest Physicians. Epidemiology, mechanisms, and risks: American College of Chest Physicians guidelines for the prevention and management of postoperative atrial fibrillation after cardiac surgery. Chest. 2005 Aug;128(2 Suppl):9S-16S. doi: 10.1378/chest.128.2_suppl.9s. PMID 16167659
- [Background] Chew JT, Ong KK. Atrial arrhythmias post coronary bypass grafting. Singapore Med J. 1993 Oct;34(5):430-4. PMID 8153692
- [Background] Alexander KP, Peterson ED. Coronary artery bypass grafting in the elderly. Am Heart J. 1997 Nov;134(5 Pt 1):856-64. doi: 10.1016/s0002-8703(97)80008-7. No abstract available. PMID 9398097
- [Background] Ad N, Snir E, Vidne BA, Golomb E. Histologic atrial myolysis is associated with atrial fibrillation after cardiac operation. Ann Thorac Surg. 2001 Sep;72(3):688-93. doi: 10.1016/s0003-4975(01)02882-x. PMID 11565642
- [Background] Ak K, Akgun S, Tecimer T, Isbir CS, Civelek A, Tekeli A, Arsan S, Cobanoglu A. Determination of histopathologic risk factors for postoperative atrial fibrillation in cardiac surgery. Ann Thorac Surg. 2005 Jun;79(6):1970-5. doi: 10.1016/j.athoracsur.2004.12.029. PMID 15919294
- [Background] Goette A, Juenemann G, Peters B, Klein HU, Roessner A, Huth C, Rocken C. Determinants and consequences of atrial fibrosis in patients undergoing open heart surgery. Cardiovasc Res. 2002 May;54(2):390-6. doi: 10.1016/s0008-6363(02)00251-1. PMID 12062343
- [Background] Serri K, Reant P, Lafitte M, Berhouet M, Le Bouffos V, Roudaut R, Lafitte S. Global and regional myocardial function quantification by two-dimensional strain: application in hypertrophic cardiomyopathy. J Am Coll Cardiol. 2006 Mar 21;47(6):1175-81. doi: 10.1016/j.jacc.2005.10.061. Epub 2006 Feb 23. PMID 16545649
- [Background] Richand V, Lafitte S, Reant P, Serri K, Lafitte M, Brette S, Kerouani A, Chalabi H, Dos Santos P, Douard H, Roudaut R. An ultrasound speckle tracking (two-dimensional strain) analysis of myocardial deformation in professional soccer players compared with healthy subjects and hypertrophic cardiomyopathy. Am J Cardiol. 2007 Jul 1;100(1):128-32. doi: 10.1016/j.amjcard.2007.02.063. Epub 2007 May 21. PMID 17599454
- [Background] Weidemann F, Niemann M, Herrmann S, Kung M, Stork S, Waller C, Beer M, Breunig F, Wanner C, Voelker W, Ertl G, Bijnens B, Strotmann JM. A new echocardiographic approach for the detection of non-ischaemic fibrosis in hypertrophic myocardium. Eur Heart J. 2007 Dec;28(24):3020-6. doi: 10.1093/eurheartj/ehm454. Epub 2007 Nov 1. PMID 17981828
- [Background] Park TH, Nagueh SF, Khoury DS, Kopelen HA, Akrivakis S, Nasser K, Ren G, Frangogiannis NG. Impact of myocardial structure and function postinfarction on diastolic strain measurements: implications for assessment of myocardial viability. Am J Physiol Heart Circ Physiol. 2006 Feb;290(2):H724-31. doi: 10.1152/ajpheart.00714.2005. Epub 2005 Sep 23. PMID 16183729
- [Background] Verma A, Wazni OM, Marrouche NF, Martin DO, Kilicaslan F, Minor S, Schweikert RA, Saliba W, Cummings J, Burkhardt JD, Bhargava M, Belden WA, Abdul-Karim A, Natale A. Pre-existent left atrial scarring in patients undergoing pulmonary vein antrum isolation: an independent predictor of procedural failure. J Am Coll Cardiol. 2005 Jan 18;45(2):285-92. doi: 10.1016/j.jacc.2004.10.035. PMID 15653029
- [Background] Hwang HJ, Choi EY, Rhee SJ, Joung B, Lee BH, Lee SH, Kim J, Lee MH, Jang Y, Chung N, Kim SS. Left atrial strain as predictor of successful outcomes in catheter ablation for atrial fibrillation: a two-dimensional myocardial imaging study. J Interv Card Electrophysiol. 2009 Nov;26(2):127-32. doi: 10.1007/s10840-009-9410-y. Epub 2009 Jun 16. PMID 19529886
- [Background] Di Salvo G, Caso P, Lo Piccolo R, Fusco A, Martiniello AR, Russo MG, D'Onofrio A, Severino S, Calabro P, Pacileo G, Mininni N, Calabro R. Atrial myocardial deformation properties predict maintenance of sinus rhythm after external cardioversion of recent-onset lone atrial fibrillation: a color Doppler myocardial imaging and transthoracic and transesophageal echocardiographic study. Circulation. 2005 Jul 19;112(3):387-95. doi: 10.1161/CIRCULATIONAHA.104.463125. Epub 2005 Jul 8. PMID 16006491
- [Background] Kuppahally SS, Akoum N, Burgon NS, Badger TJ, Kholmovski EG, Vijayakumar S, Rao SN, Blauer J, Fish EN, Dibella EV, Macleod RS, McGann C, Litwin SE, Marrouche NF. Left atrial strain and strain rate in patients with paroxysmal and persistent atrial fibrillation: relationship to left atrial structural remodeling detected by delayed-enhancement MRI. Circ Cardiovasc Imaging. 2010 May;3(3):231-9. doi: 10.1161/CIRCIMAGING.109.865683. Epub 2010 Feb 4. PMID 20133512
- [Background] Anne W, Willems R, Roskams T, Sergeant P, Herijgers P, Holemans P, Ector H, Heidbuchel H. Matrix metalloproteinases and atrial remodeling in patients with mitral valve disease and atrial fibrillation. Cardiovasc Res. 2005 Sep 1;67(4):655-66. doi: 10.1016/j.cardiores.2005.04.016. PMID 15913581
- [Background] Ware JS, Petretto E, Cook SA. Integrative genomics in cardiovascular medicine. Cardiovasc Res. 2013 Mar 15;97(4):623-30. doi: 10.1093/cvr/cvs303. Epub 2012 Sep 27. PMID 23024270
- [Background] Heinig M, Petretto E, Wallace C, Bottolo L, Rotival M, Lu H, Li Y, Sarwar R, Langley SR, Bauerfeind A, Hummel O, Lee YA, Paskas S, Rintisch C, Saar K, Cooper J, Buchan R, Gray EE, Cyster JG; Cardiogenics Consortium; Erdmann J, Hengstenberg C, Maouche S, Ouwehand WH, Rice CM, Samani NJ, Schunkert H, Goodall AH, Schulz H, Roider HG, Vingron M, Blankenberg S, Munzel T, Zeller T, Szymczak S, Ziegler A, Tiret L, Smyth DJ, Pravenec M, Aitman TJ, Cambien F, Clayton D, Todd JA, Hubner N, Cook SA. A trans-acting locus regulates an anti-viral expression network and type 1 diabetes risk. Nature. 2010 Sep 23;467(7314):460-4. doi: 10.1038/nature09386. Epub 2010 Sep 8. PMID 20827270
- [Background] Petretto E, Sarwar R, Grieve I, Lu H, Kumaran MK, Muckett PJ, Mangion J, Schroen B, Benson M, Punjabi PP, Prasad SK, Pennell DJ, Kiesewetter C, Tasheva ES, Corpuz LM, Webb MD, Conrad GW, Kurtz TW, Kren V, Fischer J, Hubner N, Pinto YM, Pravenec M, Aitman TJ, Cook SA. Integrated genomic approaches implicate osteoglycin (Ogn) in the regulation of left ventricular mass. Nat Genet. 2008 May;40(5):546-52. doi: 10.1038/ng.134. PMID 18443592